CLINICAL TRIAL: NCT01632059
Title: Examination of ADMA (Asymmetric-dimethylarginine)-Serum Level and DDAH II (Dimethylarginine Dimethylaminohydrolase)- Polymorphism in Patients With Severe Sepsis and Septic Shock as Prognostic Value
Brief Title: Examination of ADMA Serum Level and DDAH II
Acronym: ADSeS
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: ADSeS (PV3927)
Record Dates: First submitted 2012-03-13; First posted 2012-06-29 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Septic Shock; Sepsis
Keywords: ADMA; DDAH II; SAPS; SOFA; Sepsis; Procalcitonin; ICU; mortality; length of stay
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- septical patients: inclusion criteria are severe sepsis and septical shock and must be > 18 y/o

SUMMARY:
Examination of ADMA (Asymmetric-Dimethylarginine)-serum level and DDAH II (Dimethylarginine Dimethylaminohydrolase)- Polymorphism in patients with severe Sepsis and septic shock as prognostic value.

This study looks into ADMA as a good prognostic factor for sepsis. Further more the dependency of the ADMA level to the DDAH II polymorphisms is reviewed this study.

DETAILED DESCRIPTION:
Secondary targets are the mortality (28 days ICU), the length of hospitalisation in ICU and peripheral station, the severity of the illness (SAPS II score), the SOFA-score values in the progress and the procalcitonin values in the progress

ELIGIBILITY:
Inclusion Criteria:

* >18 y/o
* sepsis
* septical shock

Exclusion Criteria:

* primary cardiogenic shock
* pregnancy
* breastfeeding
* non compliance
* moribund status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 y/o with sepsis and/or septical shock
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
ADMA serum levels | 7 days
  measuring of ADMA serum levels on day 1, 3, 7

SECONDARY OUTCOMES:
28 day mortality | 28 day
hospitalisation (ICU and peripheral) | 28 days
severity of illness | 28 days
DDAH Ii polymorphism | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, Priv.-Doz., Study Director — Director of critical care center
Locations (1):
- Universitätskrankenhaus Hamburg Eppendorf, Hamburg, Germany

REFERENCES:
- See also: Related Info — http://www.uke.uni-hamburg.de